CLINICAL TRIAL: NCT01875731
Title: Efficacy of BPS (Bacterial Pneumonia Score) Guided Antibiotic Use in Children With Community Acquired Pneumonia on Reducing Antibiotic Use as Compared to Standard Care Practice (Current Guidelines for CAP) in the Era of Pneumococcal Vaccine
Brief Title: Bacterial Pneumonia Score (BPS) Guided Antibiotic Use in Children With Pneumonia and Pneumococcal Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HGNPE 67-2012
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Community Acquired Pneumonia
Keywords: Pneumonia; Acute respiratory infection; Decision-support techniques
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Guidelines as Topic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BPS (Bacterial Pneumonia Score) (Experimental): Strategy based on BPS guided antibiotic use
  Interventions: Behavioral: BPS
- Guideline (Active Comparator): Strategy based on enforced guideline guided antibiotic use
  Interventions: Behavioral: Guideline

INTERVENTIONS:
Behavioral: BPS — In this study a strategy based on BPS guided antibiotic use in children with community acquired pneumonia implementation will be compared with enforced guideline.
  Arms: BPS (Bacterial Pneumonia Score)
Behavioral: Guideline — Strategy based on enforced guideline guided antibiotic use
  Arms: Guideline

SUMMARY:
The aim of this study is to test if BPS (Bacterial Pneumonia Score) guided antibiotic use in children with non severe community acquired pneumonia (CAP) and pneumoccocal vaccine will reduce antibiotic use as compared to standard care practice (current guidelines for CAP).

DETAILED DESCRIPTION:
Background: Pneumonia is a leading cause of mortality in children. Despite more than 50% of pneumonias are due to viruses, because it is difficult to rule out bacterial etiology, initial management of pneumonia in children usually includes antibiotics, often unnecessary. In 2006 was designed and validated a clinical prediction rule (BPS: Bacterial Pneumonia Score) which accurately identifies hospitalized children's risk of bacterial pneumonia. Recently, we assessed BPS efficacy on reducing antibiotic use by 50% in children with CAP, in an ambulatory setting. However, BPS was tested in children not vaccinated against S. pneumoniae.

Aim: The aim of this study is to test if BPS guided antibiotic use in children with non severe community acquired pneumonia will reduce antibiotic use as compared to standard care practice (current guidelines for CAP)in children vaccinated against S. penumoniae.

Design: This is a randomized, controlled, blinded trial, to assess antibiotics use regarding two methods for initial management of children aged 3-60 months with non severe community acquired pneumonia and pneumoccocal vaccine. Children will be randomly allocate to be managed according to BPS or currently enforced guidelines. Use of antibiotics (%) and clinical outcome of both groups will be compared.

Setting: Tertiary children hospital in Buenos Aires, Argentina. Patients: Consecutive children aged 3-60 months assisted for non severe community acquired pneumonia as outpatients. Patients with wheezing, severe pneumonia, pulmonary or cardiovascular chronic disease, or antibiotic use or hospitalization in the previous two weeks will be excluded.

Endpoints:

Primary: Use of antibiotics in each group (proportion) Secondary: Treatment failure (proportion) in each group Endpoints will be assessed at baseline and after 1, 2, 5, 7 and 10 days by a blinded investigator.

Intervention: Patients with CAP will be randomized (1:1) to BPS versus enforced guidelines. In the BPS group antibiotics will be indicated in patients with a BPS ≥ 4 points, while in the control group antibiotics will be indicated according to current guidelines.

Variables and measurement: Antibiotic use will be defined as initial use of any antibiotic, immediately after diagnosis. Treatment failure will be defined as persistence of fever after 2 days, or tachypnea or diminishing in respiratory rate less than 5 bpm. after 2 days, or signs of severe pneumonia or requiring or changing antibiotics at any time.

Study hypothesis: BPS antibiotic use guidance will reduce at least 20% antibiotic use, as compared to standard care practice.

Analyses: These will be done based on an intention-to-treat and a per-protocol principle. With an assumed 20% less use of antibiotics in the intervention group, a maximum of 5% losses to follow-up, a confidence of 5% and power of 90%, the total sample size is 60. This will allow detecting a difference in clinical outcome of 28%. Proportion will be compared by Chi square test.

Interim monitoring: Regular review of serious adverse events, quality and integrity of the study by an independent data safety and monitoring board. Safety interim analysis after 50% of the patients recruited.

Significance: Due to the high prevalence of CAP in children, this study will offer the potential for a substantial reduction in health costs and antibiotics resistance.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-60 months assisted as outpatients for non severe community acquired pneumonia and pneumoccocal vaccine and complete immunisation with pneumoccocal vaccine.

Exclusion Criteria:

* Wheezing
* Severe pneumonia
* Pulmonary or cardiovascular chronic disease
* Antibiotic use in the previous two weeks
* Hospitalization for any reason in the previous two weeks

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando A Torres, MD, PhD, Principal Investigator — Hospital de Niños Pedro de Elizalde
Locations (1):
- Hospital General de NIños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno L, Krishnan JA, Duran P, Ferrero F. Development and validation of a clinical prediction rule to distinguish bacterial from viral pneumonia in children. Pediatr Pulmonol. 2006 Apr;41(4):331-7. doi: 10.1002/ppul.20364. PMID 16493666
- [Background] Ferrero F, Torres F, Noguerol E, Gonzalez N, Lonegro L, Chiolo MJ, Ossorio MF, Benguigui Y. [Evaluation of two standardized methods for chest radiographs interpretation in children with pneumonia]. Arch Argent Pediatr. 2008 Dec;106(6):510-4. doi: 10.1590/S0325-00752008000600007. Spanish. PMID 19107303

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BPS (Bacterial Pneumonia Score) | Guideline
Started | 34 | 32
Completed | 33 | 32
Not Completed | 1 | 0
Not completed — Fail to obtain lab sample | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BPS (Bacterial Pneumonia Score) | Guideline | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: months] | 17.2 (10.2) | 17.5 (11) | 17.5 (10.8)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 19 | 14 | 33
Region of Enrollment [Number; unit: participants]
  Argentina | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Use of Antibiotics in Each Group
Description: Number of participants with use of any antibiotic, at any time after diagnosis
Time Frame: At day 7 from baseline
Measure: Number; unit: participants
Arm/Group | BPS (Bacterial Pneumonia Score) | Guideline
Number analyzed (Participants) | 33 | 32
participants | 9 | 21
Statistical Analysis 1: Comparison: BPS (Bacterial Pneumonia Score) vs Guideline; Test type: Superiority or Other; p = 0.01, Chi-squared; Odds Ratio (OR) = 5.09, 95% CI 2-sided [1.57 to 16.8]

2. Secondary Outcome: Treatment Failure in Each Group
Description: Number of participants with persistence of fever after 2 days, or tachypnea or diminishing in respiratory rate less than 5 bpm. after 2 days, or signs of severe pneumonia or requiring or changing antibiotics at any time.
Time Frame: 1, 2, 5, 7 and 10 days from baseline
Measure: Number; unit: participants
Arm/Group | BPS (Bacterial Pneumonia Score) | Guideline
Number analyzed (Participants) | 33 | 32
participants | 3 | 4
Statistical Analysis 1: Comparison: BPS (Bacterial Pneumonia Score) vs Guideline; Test type: Superiority or Other; p = 0.71, Chi-squared; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.1 to 4.09]

ADVERSE EVENTS:
Arm/Group | BPS (Bacterial Pneumonia Score) | Guideline
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes